CLINICAL TRIAL: NCT01715415
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of ABT450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 Co-administered With Ribavirin (RBV) in Treatment-Experienced Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection (SAPPHIRE-II)
Brief Title: A Study to Evaluate Chronic Hepatitis C Infection in Treatment Experienced Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-098; 2012-002035-29 (EudraCT Number)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C; Treatment-Experienced; Null responder; Partial Responder; Chronic Hepatitis; Hepatitis C Genotype 1; Interferon-Free; Hepatitis C Virus; Relapser; Non responder; Viekira Pak; ombitasvir; ribavirin; ritonavir; paritaprevir; dasabuvir
MeSH Terms: conditions — Hepatitis C; Hepatitis, Chronic | interventions — dasabuvir; ombitasvir; paritaprevir; Viekira Pak; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABT-450/r/ABT-267 and ABT-333, plus RBV (Experimental): Double-blind ABT-450/r/ABT-267 (150 mg/100 mg/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based ribavirin (RBV; dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin
- Placebo Followed by ABT-450/r/ABT-267 and ABT-333, plus RBV (Experimental): Double-blind placebo for 12 weeks, followed by open-label ABT-450/r/ABT-267 (150 mg/100 mg/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (RBV; dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin; Drug: Placebo for ABT-450/r/ABT-267; Drug: Placebo for ABT-333; Drug: Placebo for ribavirin

INTERVENTIONS:
Drug: ABT-450/r/ABT-267, ABT-333 — Tablet; ABT-450 coformulated with ritonavir and ABT-267, ABT-333 tablet
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ABT-333 also known as dasabuvir; Viekira PAK
Drug: Ribavirin — Capsule (double-blind treatment period), tablet (open-label treatment period)
Drug: Placebo for ABT-450/r/ABT-267 — Tablet
  Arms: Placebo Followed by ABT-450/r/ABT-267 and ABT-333, plus RBV
Drug: Placebo for ABT-333 — Tablet
  Arms: Placebo Followed by ABT-450/r/ABT-267 and ABT-333, plus RBV
Drug: Placebo for ribavirin — Capsule
  Arms: Placebo Followed by ABT-450/r/ABT-267 and ABT-333, plus RBV

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ABT-450, ritonavir and ABT-267 (ABT-450/r/ABT-267; ABT-267 also known as ombitasvir) and ABT-333 (also known as dasabuvir) co-administered with ribavirin (RBV) in hepatitis C virus genotype 1 infected treatment-experienced adults.

ELIGIBILITY:
Inclusion Criteria:

* Females must be post-menopausal for at least 2 years or surgically sterile or practicing specific forms of birth control.
* Chronic hepatitis C, genotype 1 infection and HCV RNA level greater than 10,000 IU/mL at screening.
* Previous treatment failure of peg-interferon and ribavirin (pegIFN and RBV).
* No evidence of liver cirrhosis.

Exclusion Criteria:

* Positive screen for drugs or alcohol.
* Significant sensitivity to any drug.
* Use of contraindicated medications within 2 weeks of dosing.
* Certain predefined abnormal laboratory tests.
* Positive hepatitis B surface antigen or anti-human immunodeficiency virus antibody.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Enejosa, MD, Study Director — AbbVie

REFERENCES:
- [Result] Zeuzem S, Jacobson IM, Baykal T, Marinho RT, Poordad F, Bourliere M, Sulkowski MS, Wedemeyer H, Tam E, Desmond P, Jensen DM, Di Bisceglie AM, Varunok P, Hassanein T, Xiong J, Pilot-Matias T, DaSilva-Tillmann B, Larsen L, Podsadecki T, Bernstein B. Retreatment of HCV with ABT-450/r-ombitasvir and dasabuvir with ribavirin. N Engl J Med. 2014 Apr 24;370(17):1604-14. doi: 10.1056/NEJMoa1401561. Epub 2014 Apr 10. PMID 24720679
- [Derived] Feld JJ, Bernstein DE, Younes Z, Vlierberghe HV, Larsen L, Tatsch F, Ferenci P. Ribavirin dose management in HCV patients receiving ombitasvir/paritaprevir/ritonavir and dasabuvir with ribavirin. Liver Int. 2018 Sep;38(9):1571-1575. doi: 10.1111/liv.13708. Epub 2018 Mar 14. PMID 29377566
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- ABT-450/r/ABT-267 and ABT-333, Plus RBV: Double-blind ABT-450/r/ABT-267 (150 mg/100 mg/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based ribavirin (RBV; dosed 1,000 to 1,200 mg/day divided twice daily) for 12 weeks
- Placebo Followed by ABT-450/r/ABT-267 and ABT-333, Plus RBV: Double-blind placebo for 12 weeks, followed by open-label ABT-450/r/ABT-267 (150 mg/100 mg/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (RBV; dosed 1,000 to 1,200 mg/day divided twice daily) for 12 weeks
Period: Double-blind Treatment
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | Placebo Followed by ABT-450/r/ABT-267 and ABT-333, Plus RBV
Started | 297 | 98
Randomized But Not Treated | 0 | 1
Completed | 292 (The number of participants who completed double-blind study drug.) | 96 (The number of participants who completed double-blind study drug.)
Not Completed | 5 | 2
Not completed — Did Not Receive Study Drug | 0 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 0
Period: Open-label Treatment
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | Placebo Followed by ABT-450/r/ABT-267 and ABT-333, Plus RBV
Started | 0 (not applicable to this arm) | 96
Completed | 0 (not applicable to this arm) | 94 (The number of participants who completed open-label study drug.)
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Subject Noncompliant | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all randomized participants who received at least 1 dose of blinded study drug.
Groups:
- Placebo: Double-blind placebo for 12 weeks
- Total: Total of all reporting groups
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | Placebo | Total
Number analyzed (Participants) | 297 | 97 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.26) | 54.9 (8.46) | 52.5 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 37 | 167
  Male | 167 | 60 | 227

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of active study drug
Population: Intent-to-treat (ITT) Population: All randomized participants who received at least 1 dose of blinded study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 297
percentage of participants | 96.3
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV; With a sample size of 300 subjects and assuming that 85% of the subjects in Arm A will achieve sustained virologic response (SVR) 12, this study has greater than 90% power to demonstrate non-inferiority with a 2-sided 95% lower confidence bound greater than 60% and greater than 90% power to demonstrate superiority with a 2-sided 95% lower confidence bound greater than 70% (based on the normal approximation of a single binomial proportion); Test type: Non-Inferiority or Equivalence — Based on historical SVR rates for noncirrhotic peg-interferon/ribavirin (pegIFN/RBV) treatment-experienced subjects administered telaprevir plus pegIFN/RBV, the lower confidence bound (LCB) of the 95% confidence interval (CI) must have exceeded 60% to achieve noninferiority of the ABT-450/r/ABT-267 and ABT-333, plus RBV treatment group as compared with the historical rate for telaprevir plus pegIFN and RBV, and the LCB of the 95% CI must have exceeded 70% to achieve superiority; Percentage of Participants with SVR12 = 96.3, 95% CI 2-sided [94.1 to 98.4] — 95% CI calculated using the normal approximation to the binomial distribution. In order to control the Type I error rate at 0.05, a fixed-sequence testing procedure was used to proceed through the primary and numbered secondary efficacy endpoints

2. Secondary Outcome: Percentage of Participants With Normalization of Alanine Aminotransferase (ALT) at Final Treatment Visit During the Double-Blind Treatment Period
Description: Normalization is defined as alanine aminotransferase less than or equal to the upper limit of normal (ULN) at final treatment visit for participants with alanine aminotransferase greater than ULN at baseline.
Time Frame: At 12 weeks
Population: Intent-to-treat (ITT) Population: All randomized participants who received at least 1 dose of blinded study drug and had ALT ≥ ULN of the reference range at baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV | Placebo
Number analyzed (Participants) | 224 | 78
percentage of participants | 96.9 | 12.8
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — In order to control the Type I error rate at 0.05, a fixed-sequence testing procedure will be used to proceed through the primary and the first 3 secondary endpoints in the order numbered below

3. Secondary Outcome: Percentage of HCV Genotype 1a-infected Participants With Sustained Virologic Response 12 Weeks After Treatment
Description: as for outcome 1
Time Frame: 12 weeks after the last actual dose of active study drug
Population: Intent-to-treat (ITT) Population: All randomized participants in the Double-blind ABT-450/r/ABT-267 and ABT-333, plus RBV treatment arm with HCV genotype 1a who received at least 1 dose of blinded study drug. 1 participant, who had genotype 1 HCV with an indeterminate subgenotype, is not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 173
percentage of participants | 96.0
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV; Test type: Non-Inferiority or Equivalence — Based on historical SVR rates for noncirrhotic pegIFN/RBV treatment-experienced subjects of the appropriate HCV genotype 1 subtype administered telaprevir plus pegIFN/RBV, the lower confidence bound (LCB) of the 95% confidence interval (CI) must have exceeded 65% to achieve superiority of the ABT-450/r/ABT-267 and ABT-333, plus RBV treatment group as compared with the historical rate for telaprevir plus pegIFN and RBV; Percentage of Participants with SVR12 = 96.0, 95% CI 2-sided [93.0 to 98.9] — 95% CI calculated using the normal approximation to the binomial distribution

4. Secondary Outcome: Percentage of HCV Genotype 1b-infected Participants With Sustained Virologic Response 12 Weeks After Treatment
Description: as for outcome 1
Time Frame: 12 weeks after the last actual dose of active study drug
Population: Intent-to-treat (ITT) Population: All randomized participants in the Double-blind ABT-450/r/ABT-267 and ABT-333, plus RBV treatment arm with HCV genotype 1b who received at least 1 dose of blinded study drug. 1 participant, who had genotype 1 HCV with an indeterminate subgenotype, is not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 123
percentage of participants | 96.7
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 and ABT-333, Plus RBV; Test type: Non-Inferiority or Equivalence — Based on historical SVR rates for noncirrhotic pegIFN/RBV treatment-experienced subjects of the appropriate HCV genotype 1 subtype administered telaprevir plus pegIFN/RBV, the lower confidence bound (LCB) of the 95% confidence interval (CI) must have exceeded 77% to achieve superiority of the ABT-450/r/ABT-267 and ABT-333, plus RBV treatment group as compared with the historical rate for telaprevir plus pegIFN and RBV; Percentage of Participants with SVR12 = 96.7, 95% CI 2-sided [93.6 to 99.9]

5. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure During the Double-blind Treatment Period: ABT-450/r/ABT-267 and ABT-333, Plus RBV Arm
Description: Virologic failure was defined as rebound (hepatitis C virus ribonucleic acid [HCV RNA] ≥ lower limit of quantification [LLOQ] after HCV RNA < LLOQ or increase in HCV RNA of at least 1 log10 IU/mL) or failure to suppress (all on-treatment values of plasma HCV RNA ≥ LLOQ with at least 36 days of treatment) during treatment.
Time Frame: 12 weeks after the last actual dose of active study drug
Population: Intent-to-treat (ITT) Population: All randomized participants who received at least 1 dose of blinded study drug in the Double-blind ABT-450/r/ABT-267 and ABT-333, plus RBV treatment arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 297
percentage of participants | 0 [0.0 to 0.0]

6. Secondary Outcome: Percentage of Participants With Virologic Relapse After Treatment: ABT-450/r/ABT-267 and ABT-333, Plus RBV Arm
Description: Participants were considered to have virologic relapse after treatment if they had confirmed quantifiable plasma hepatitis C virus ribonucleic acid (HCV RNA) greater than or equal to the lower limit of quantification (≥ LLOQ) between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA < LLOQ at the end of treatment.
Time Frame: Within 12 weeks post-treatment
Population: Intent-to-treat (ITT) Population: All randomized participants who received at least 1 dose of blinded study drug with HCV RNA < LLOQ at the final treatment visit who completed treatment in the Double-blind ABT-450/r/ABT-267 and ABT-333, plus RBV treatment arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 and ABT-333, Plus RBV
Number analyzed (Participants) | 293
percentage of participants | 2.4 [0.6 to 4.1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the start of active study drug administration (double-blind [DB] or open-label [OL] active) to 30 days after the last dose of active study drug (total 16 weeks).
Description: DB Placebo Arm: AEs collected from start of placebo until 30 days following discontinuation of placebo and prior to the OL period (if applicable; total 16 weeks). Serious AES collected from informed consent until the end of participation in the study (12 weeks, DB period; 12 weeks, OL period + 48-week post-treatment period; total up to 72 weeks).
Groups:
- Double Blind ABT-450/r/ABT-267 and ABT-333, Plus RBV: Double-blind ABT-450/r/ABT-267 (150 mg/100 mg/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based ribavirin (RBV; dosed 1,000 to 1,200 mg/day divided twice daily) for 12 weeks
- Double Blind Placebo: Double-blind placebo for 12 weeks
- Open Label ABT-450/r/ABT-267 and ABT-333, Plus RBV: Open-label ABT-450/r/ABT-267 (150 mg/100 mg/25 mg once daily) and ABT-333 (250 mg twice daily), plus weight-based RBV (RBV; dosed 1,000 to 1,200 mg/day divided twice daily) for 12 weeks
Arm/Group | Double Blind ABT-450/r/ABT-267 and ABT-333, Plus RBV | Double Blind Placebo | Open Label ABT-450/r/ABT-267 and ABT-333, Plus RBV
Serious Adverse Events (participants affected / at risk) | 6/297 | 1/97 | 3/96
Other Adverse Events (participants affected / at risk) | 254/297 | 74/97 | 74/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=297) | Double Blind Placebo (N=97) | Open Label ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=96)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=297) | Double Blind Placebo (N=97) | Open Label ABT-450/r/ABT-267 and ABT-333, Plus RBV (N=96)
ANAEMIA (Blood and lymphatic system disorders) | 16 | 0 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 16 | 6 | 9
CONSTIPATION (Gastrointestinal disorders) | 4 | 6 | 0
DIARRHOEA (Gastrointestinal disorders) | 39 | 12 | 8
DYSPEPSIA (Gastrointestinal disorders) | 18 | 3 | 7
NAUSEA (Gastrointestinal disorders) | 59 | 17 | 13
VOMITING (Gastrointestinal disorders) | 19 | 0 | 3
ASTHENIA (General disorders) | 47 | 11 | 13
FATIGUE (General disorders) | 99 | 22 | 16
IRRITABILITY (General disorders) | 16 | 8 | 6
NASOPHARYNGITIS (Infections and infestations) | 21 | 5 | 8
DECREASED APPETITE (Metabolism and nutrition disorders) | 20 | 2 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 19 | 7 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 | 3 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 23 | 10 | 5
DIZZINESS (Nervous system disorders) | 25 | 5 | 5
DYSGEUSIA (Nervous system disorders) | 10 | 5 | 3
HEADACHE (Nervous system disorders) | 108 | 34 | 18
ANXIETY (Psychiatric disorders) | 14 | 4 | 7
DEPRESSED MOOD (Psychiatric disorders) | 5 | 5 | 1
INSOMNIA (Psychiatric disorders) | 42 | 7 | 10
COUGH (Respiratory, thoracic and mediastinal disorders) | 32 | 5 | 11
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 37 | 10 | 13
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 8
DRY SKIN (Skin and subcutaneous tissue disorders) | 22 | 3 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 41 | 5 | 12
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 11 | 5 | 3
RASH (Skin and subcutaneous tissue disorders) | 26 | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.